CLINICAL TRIAL: NCT01926717
Title: A Comparative Clinical Research on Single Roux-en-Y and Traditional Roux-en-Y of Pancreaticojejunostomy-choledochojejunostomy For Treatment of Obstruction of Pancreatic Duct and Bile Duct
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chengyi Sun (Other)
Responsible Party: Sponsor-Investigator, Chengyi Sun, Department of Hepatobiliary Surgery, The First Affiliated Hospital of Guangzhou Medical University
Organization: The First Affiliated Hospital of Guangzhou Medical University (Other)
Other Study IDs: GYGDWK-02
Record Dates: First submitted 2013-08-19; First posted 2013-08-21 (Estimated); Last update posted 2016-03-08 (Estimated); Status verified 2016-03

CONDITIONS: Pancreatic Cancer
Keywords: Single Roux-y of Pancreaticojejunostomy-choledochojejunostomy
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Single Roux-y of Pancreaticojejunostomy-choledochojejunostomy
- Pancreaticoduodenectomy

SUMMARY:
This study is being done to learn more about how different surgery procedures bring back the quality of life.After removing the small intestine at least 20cm in patients with pancreatic cancer, Some patients develop problems because they are disorder their digestive system, such as cramping, heartburn,vomiting.

ELIGIBILITY:
Inclusion Criteria:

* Patient 30 years of age or older
* Pathologically confirmed pancreatic cancer (biopsy may be performed at our institution)
* No evidence of metastases(a)
* decide performe Roux-en-Y(b)
* single Roux-en-Y reconstruction is technically feasible(c)
* Patients will be registered and consent obtained, if the surgeon believes there is no evidence of metastases. If metastatic disease is identified at the time of operation, the patient will not be randomized.
* Patients will be conditionally enrolled, and consent obtained, if the surgeon believes the patient may need a sngle Roux-en-Y at the time of operation. If a sngle Roux-en-Y is not performed, the patient will not be randomized.
* the surgeon feels that the single Roux-en-Y is not technically feasible at the time of operation,the patients will be excluded. This may be due to prior abdominal surgery, anatomic variants, or anything else at the surgeon's discretion.

Exclusion Criteria:

* Not expected to be able to provide follow-up over 2 years (due to geographic or other limitations)

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with pancreatic cancer
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2010-12; Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
The secretion function of the pancreas | Participants will be followed for overall 3 year after surgery

SECONDARY OUTCOMES:
The function of biliary tract | Participants will be followed for overall 3 year after surgery

OTHER OUTCOMES:
The relief of abdominal pain symptom | Participants will be followed for overall 3 year after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- The Affiliated Hospital of Guiyang Medical College, Guiyang, Guizhou, China